CLINICAL TRIAL: NCT04575623
Title: Central Auditory and Cognitive Functions in Patients Suffering From Migraine
Brief Title: Auditory Functions in Patients With Migraine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Weaam Noaman Mohamed Aziz Aldin, Principal investigator, Assiut University
Other Study IDs: Patients with migraine
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: It will consist of 120 patients suffering from migraine according to international classification of headache
  Interventions: Diagnostic Test: Duration Pattern test (DPT) /Dichotic Digits Test (DDT) /Auditory fusion test-revised (ART-R)/; Device: Dual band pure tone audiometer (Orbiter 992). -Impedance audiometer (AT 235h). -Sound treated booth (industrial acoustic company IAC model 1602-A-t) -Panasonic stereo CD player SA-AK 240.

INTERVENTIONS:
Diagnostic Test: Duration Pattern test (DPT) /Dichotic Digits Test (DDT) /Auditory fusion test-revised (ART-R)/ — Central auditory function evaluation including:
  * Duration Pattern test (DPT) designed to test temporal ordering abilities.
  * Dichotic Digits Test (DDT) it assesses binaural integration skills.
  * Auditory fusion test-revised (ART-R) to measure temporal resolution.
  * speech in test to assess central auditory function.
Device: Dual band pure tone audiometer (Orbiter 992). -Impedance audiometer (AT 235h). -Sound treated booth (industrial acoustic company IAC model 1602-A-t) -Panasonic stereo CD player SA-AK 240. — Cognitive function evaluation including:
  -Recording of event-related potentials (ERPs) by using odd ball paradigm auditoryP300 wave in evaluating cerebral information processing.
  Equipment:
  * Dual band pure tone audiometer (Orbiter 992).
  * Impedance audiometer (AT 235h).
  * Sound treated booth (industrial acoustic company IAC model 1602-A-t)
  * Panasonic stereo CD player SA-AK 240.

SUMMARY:
Migraine is a neurological disease associated with an altered cortical excitability level . The prevalence of migraine is10.5% of adults in Assiut governorate, and is more frequent in women and in individuals with higher education level . There is evidence that migraine patients could present cognitive deficits, being the affected functions memory, processing information speed and attention. It was found that the prevalence of migraine in AlQuseir was 4.8/100 and the highest figures found during early adult life(18-40) years old .Patients with migraine found to perform significantly worse in duration pattern test(DPT),non-verbal dichotic test ,speech in noise (SPIN)test and found to have longer p300 frequency stimulus latency which indicate presence of cognitive and central auditory processing dysfunction

DETAILED DESCRIPTION:
The definition of central auditory processing CAP is based on auditory functions . Central auditory processing CAP involves a large number of skills which are highly dependent on a set integrity of the auditory pathways, from the outer ear to the auditory cortex. These skills include auditory selective attention, sound detection, and localization, discrimination of isolated and sequential sounds, as well as speech recognition, auditory comprehension and memory .

central auditory processing CAP is an indispensable tool for the investigation of the function of the central nervous system . The impairment of auditory processing could cause difficulties in complex listening situations, such as understanding speech in back-ground noise, rapid or degraded speech, and problems with comprehending verbal instructions.

Central auditory perception (CAP) can be assessed by Behavioral tests, which demonstrate good correlations with electrophysiological measures . Recording of event-related potentials (ERPs), because of its objectivity and noninvasive characteristics, presents one of the most useful tools in investigating neural substrates and cerebral regions involved in specific cognitive function. It implies recording of brain activity during a cognitive task .

Among the components of ERPs, theP300 is undoubtedly the most studied cerebral wave in evaluating cerebral information processing during the course of various neurological diseases because of its easy recording and reliability . The P300 develops if the subject is actively engaged in the task of detecting the targets.

Amplitude of the wave varies with the improbability of the targets and latency with the difficulty of discriminating the target stimulus from the standard stimuli . Typical peak latency P300 latency reflects timing of mental processes and the increase of latency represents prolongation of the processing time

ELIGIBILITY:
Inclusion Criteria:

* It will consist of 100 patients suffering from migraine according to international classification of headache.
* Their age range from (18-40) years old which considered the most common affected age group ,
* Both sexes will be included.
* The study group will be further classified into two main categories migraine with and without aura.

Exclusion Criteria:

* Patients with history of systemic, neurologic or psychiatric illness.
* Patients with other types of headache.
* Patients with hearing loss.
* Patients with history of head trauma, surgery or ototoxic drug therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with migraine as study group and normal people as control group
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Determination of central auditory processing in patients with migraine | One year
  Evaluation of auditory functions in patients with migraine by using
  Duration Pattern test (DPT) designed to test temporal ordering abilities. Dichotic Digits Test (DDT) it assesses binaural integration skills. Auditory fusion test-revised (ART-R) to measure temporal resolution. speech in test to assess central auditory function.
Determination of cognitive functions in patients with migraine | One year
  Evaluation of cognitive functions in patients with migraine by Recording of event-related potentials (ERPs) by using odd ball paradigm auditoryP300 wave in evaluating cerebral information processing